CLINICAL TRIAL: NCT00572520
Title: Treating Co-morbid Obesity and Major Depressive Disorder
Brief Title: Effectiveness of Behavioral Treatments for Obesity and Major Depression in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH078012 (NIH); R01MH078012 (NIH); DAHBR 96-BHB
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Depression; Obesity
Keywords: Depressive Disorder; Weight Loss; Behavioral Treatment; Behavior Therapy; Randomized Clinical Trial
MeSH Terms: conditions — Depression; Obesity; Depressive Disorder; Weight Loss | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Evidence-based behavioral weight loss treatment with health education counseling
  Interventions: Behavioral: Weight loss treatment; Behavioral: Health education counseling
- 2 (Experimental): Evidence-based behavioral weight loss treatment with brief behavior therapy for depression
  Interventions: Behavioral: Weight loss treatment; Behavioral: Behavior therapy for depression

INTERVENTIONS:
Behavioral: Weight loss treatment — Over 2 years, this treatment involves a total of 26 group visits and 10 individual visits with a health education counselor. Group visits, led by a registered dietitian and a licensed exercise physiologist, will target diet and physical activity.
Behavioral: Behavior therapy for depression — Behavior therapy for depression will be delivered by a trained behavior therapist. Participants receiving behavioral counseling will learn about depression, links between activity and mood, and will be asked to keep a diary of moods and activities.
  Arms: 2
Behavioral: Health education counseling — Health education counseling will be delivered by a trained health education counselor. Participants receiving health education will learn about women's health topics and receive tips on staying healthy and preventing disease.
  Arms: 1

SUMMARY:
This study will compare the effectiveness of two weight loss programs, one supplemented with health education and the other supplemented with behavioral counseling, in treating women who are depressed and overweight.

DETAILED DESCRIPTION:
Obesity is one of the most alarming current health problems in the United States, with 31% percent of the population considered obese. Previous studies have shown that there is a higher incidence of depression in people who are overweight. It is not known whether depression causes obesity or vice versa, but the association may stem from the stigma of obesity or from the appetite and weight gain caused by depressive symptoms. With the increased risk of cardiovascular and other life-threatening diseases from obesity, promotion of healthful habits is important. Providing the motivational skills to adhere to these habits is also crucial, especially in people who are both overweight and depressed. This study will compare the effectiveness of two weight loss programs, one supplemented with health education and the other supplemented with behavioral counseling, in treating women who are depressed and overweight.

Participants in this 2-year study will be divided into one of two treatment groups: one group will address weight loss and depression via nutrition, exercise, and health education and the other group will address weight loss and depression via nutrition, exercise, and behavioral counseling. Participants receiving health education will learn about women's health topics and receive tips on staying healthy and preventing disease. Participants receiving behavioral counseling will learn about depression and links between activity and mood. They will also be asked to keep a diary of moods and activities. Participants in both treatment groups will undergo the same schedule of study visits and assessments. A baseline visit will include blood tests; measurements of height, weight, waist size, and blood pressure; and completion of questionnaires about depression, eating habits, and physical activity. Next, over a 3-week period, participants will receive three phone calls asking about food intake from the previous day. In the first 6 months of the study, there will be a total of 26 weekly treatment visits. These visits will consist of ten 1-hour sessions with a counselor and sixteen 90-minute sessions with a dietician. During the next 6 months, participants will continue to meet with their dieticians monthly for a total of 6 visits and will receive monthly phone calls from their counselor. Quaterly phone calls with their counselor will continue in the second year of the study. There will be three check-in appointments similar to the baseline assessment, occurring at Month 6 and Years 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for major depressive disorder
* Score of 12 to 24 on Hamilton Depression Rating Scale (HDRS)
* Body mass index (BMI) of 30 to 40 kg

Exclusion Criteria:

* Plans to move out of the area during the study
* Current smoker
* Diagnosis of bipolar disorder, a psychotic disorder, bulimia, or post-traumatic stress disorder
* Meets criteria for severe depression (HDRS score greater than 24)
* Diagnosis of type 1 or 2 diabetes
* Plans to have bariatric surgery during the study
* No access to a telephone
* Unable to walk unaided or unable to walk 1/4 mile without stopping
* Does not have written clearance from primary care physician for physical activity
* Presence of a condition that precludes dietary changes (e.g., ulcerative colitis, Crohn's disease, active diverticulitis, renal disease)
* Presence of medical conditions likely to limit lifespan
* Taking prescription weight loss medications
* Initiation of anti-depressant medication within the 3 months prior to study entry
* Taking mood stabilizers, antipsychotic medication, or medications known to affect appetite and/or weight (e.g., corticosteroids)
* Reports active suicidal ideation via SCID interview, a score of 3 on item 24 of the HDRS (active suicidal ideation), or determined to have suicidal potential by clinical staff
* Psychiatric hospitalization in the 12 months prior to study entry
* Currently receiving psychotherapy

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2007-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in body weight and the trend in body weight over time | Measured at Month 6 and Years 1 and 2

SECONDARY OUTCOMES:
Change in depression, physical activity, diet (daily caloric intake), psychosocial variables (anhedonia, exercise self-efficacy, disinhibited eating, quality of life), and cardiovascular risk factors (blood pressure, serum lipids, C-reactive protein) | Measured at Year 2
Effect of potential mediators (adherence, depression, general and physical activity, caloric intake) on weight change | Measured at Year 2

CONTACTS AND LOCATIONS:
Overall Officials: Sherry L. Pagoto, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Schneider KL, Bodenlos JS, Ma Y, Olendzki B, Oleski J, Merriam P, Crawford S, Ockene IS, Pagoto SL. Design and methods for a randomized clinical trial treating comorbid obesity and major depressive disorder. BMC Psychiatry. 2008 Sep 15;8:77. doi: 10.1186/1471-244X-8-77. PMID 18793398